CLINICAL TRIAL: NCT06086210
Title: Evaluation of the Efficacy of Low Level Laser Therapy in Ulnar Neuropathy at the Elbow in Terms of Symptoms, Clinical and Electrophysiological: A Randomized, Prospective, Double-blind Clinical Trial
Brief Title: Evaluation of the Efficacy of Low Level Laser Therapy in Ulnar Neuropathy at the Elbow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gulsah Celik (Other Government)
Responsible Party: Sponsor-Investigator, Gulsah Celik, Principal Investigator, Antalya Training and Research Hospital
Organization: Antalya Training and Research Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AntalyaTRHCelik01
Record Dates: First submitted 2023-10-07; First posted 2023-10-17 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Ulnar Nerve Entrapment at Elbow
Keywords: Low-lever laser therapy; Splint; Ulnar Nerve Entrapment at Elbow; Electroneuromyography
MeSH Terms: conditions — Cubital Tunnel Syndrome | interventions — Low-Level Light Therapy; salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: Two groups with laser treatment and sham-controlled treatment
Who Masked: Participant, Outcomes Assessor
Masking Description: Since the light coming from the probe was visible in the laser applications used in both groups, the patients were not able to learn which group they were in, meaning they were blinded. All outcome measures were evaluated by another researcher who did not know which group the patients were in, thus ensuring that the study was double-blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-level laser therapy group (Active Comparator): Low-level laser therapy was applied to the patients with the elbow at 45° flexion, creating a total of 5 areas by drawing 2 cm intervals 4 cm below the elbow and 6 cm above the elbow. The patients in the group used the elbow rest splint throughout the night during the treatment.
  Interventions: Other: Low-level laser therapy
- Sham group (Sham Comparator): Sham group was applied with a laser probe by the elbow in 45° flexion, creating a total of 5 areas by drawing 2 cm intervals 4 cm below the elbow and 6 cm above the elbow. The patients in the group used the elbow rest splint throughout the night during the treatment.
  Interventions: Other: Sham

INTERVENTIONS:
Other: Low-level laser therapy — Low-level laser therapy was applied to each area for 1 minute, with a wavelength of 808 nm and a dose of 2j/cm2 for a total of 5 minutes,10j/cm2 in continuous mode. A total of 15 sessions were applied 5 days a week for 3 weeks.
  Other Names: Medical Italia PR999 4W
  Arms: Low-level laser therapy group
Other: Sham — Sham therapy was applied to each area for 1 minute, with a wavelength of 0 nm and a dose of 0j/cm2 for a total of 5 minutes, 0j/cm2. A total of 15 sessions were applied 5 days a week for 3 weeks.
  Arms: Sham group

SUMMARY:
The purpose of this study is, to demonstrate the effectiveness of low-level laser therapy on symptoms, clinical and electrophysiological parameters in elbow ulnar neuropathy.

DETAILED DESCRIPTION:
Ulnar neuropathy of the elbow is the second most common entrapment neuropathy of the upper extremity. The ulnar nerve is prone to entrapment due to its anatomical location in the elbow. The most important cause of entrapment occurs as a result of frequent chronic mechanical compression or stretching. Repetitive flexion-extension movement of the elbow increases the pressure in both the cubital tunnel and other potential entrapment sites, causing tension in the ulnar nerve and increased intraneural pressure.

Ulnar neuropathy of the elbow, a detailed history and a comprehensive physical examination are the essential first steps in making the correct diagnosis. In case of doubt, electrophysiological studies, in particular, play an important role in diagnosis by determining both the location of nerve compression and the severity of the disease. There are conservative and surgical methods for the treatment of ulnar neuropathy in the elbow. In most patients, especially in mild and moderate entrapments, conservative treatment is preferred instead of surgery as initial treatment.

Low-level laser therapy, one of the physical therapy modalities, creates photochemical reactions and biostimulation in the cells, interstitial tissue, vascular structure and immune system. Its anti-inflammatory effect is through inhibition of Cyclooxygenase-2 enzyme and a decrease in Prostaglandin E2 levels, and its analgesic effect is by inhibiting nociceptive pathways in peripheral nerves, thus reducing pain. It has been shown to increase nerve regeneration and nerve conduction, reduce the effects of nerve compression, and may stimulate nerve healing thanks to its biophysical effect.

There is no sham-controlled study showing the effectiveness of low-level laser therapy in elbow ulnar neuropathy, the second most common entrapment neuropathy. The study was planned to investigate the effectiveness of low-level laser treatment on symptoms, clinical and electrophysiological parameters in elbow ulnar neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Ulnar neuropathy at the elbow evidenced by electrophysiological evaluation
* Symptoms onset with more than 1 months

Exclusion Criteria:

* Presence of thenar, hypothenar or intrinsic muscle atrophy,
* Diabetes mellitus
* Hypothyroidism
* Receiving an electrophysiological diagnosis of carpal tunnel syndrome, cervical radiculopathy, brachial plexopathy, thoracic outlet syndrome
* Vascular disease
* Ulnar nerve injury or trauma,
* Malignancy,
* Having received treatment for ulnar neuropathy in the elbow within the last 3 months,
* Using nonsteroidal anti-inflammatory drugs (NSAI) regularly

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | Baseline, Days 15 and Months 3
  The patient's symptoms were filled in, with the VAS score increasing from 0 to 10. The end of a 10 cm line with 0 cm indicating no complaints (best) and the end with 10 cm indicating very severe complaints (worst).

SECONDARY OUTCOMES:
Hand Grip Strength | Baseline, Days 15 and Months 3
  The hand is squeezed to grasp with maximum force, with the shoulder in adduction and neutral rotation, the elbow in 90° flexion, the forearm in midrotation and the wrist in neutral. Jamar hand dynamometer was used in measurements. Three measurements were written in kilograms (kg), with a one-minute rest between each measurement, and the average value was recorded.
Provocative Tests | Baseline, Days 15 and Months 3
  Tinel's test involves tapping the ulnar nerve in the medial epicondylar groove. In the elbow flexion test, the elbow is held in maximum flexion, the forearm is in supination, and the wrist is in full extension for 60 seconds. In the ulnar nerve compression test, the elbow is kept in 20° flexion and the forearm is kept in supination position. The examiner places his index and middle fingers over the cubital tunnel and applies pressure for 60 seconds. In all of these tests, if paresthesia or numbness occurs in the ulnar nerve distribution, the test is considered positive.
QuickDASH score | Baseline, Days 15 and Months 3
  Quick-DASH score, which quickly evaluates arm-shoulder-hand problems, consists of 11 questions. Functional evaluation of the patients' upper extremities and strains during daily living activities are questioned. The best score in total is determined as 0, and the lowest score is determined as 100.
Electrophysiological Studies | Baseline, Days 15 and Months 3
  In the electrophysiological evaluation, motor nerve conduction velocity in meter/second of the ulnar nerve at the elbow was measured.
Electrophysiological Studies | Baseline, Days 15 and Months 3
  In the electrophysiological evaluation ulnar distal latency in millisecond difference at distances measured by the centimeter method (inching) at the elbow was measured.
Electrophysiological Studies | Baseline, Days 15 and Months 3
  In the electrophysiological evaluation sensory nerve conduction velocity in meter/second at the wrist was measured.
Electrophysiological Studies | Baseline, Days 15 and Months 3
  In the electrophysiological evaluation sensory distal latency in millisecond recorded at the wrist and was measured.

CONTACTS AND LOCATIONS:
Overall Officials: Gülşah Çelik, MD, Principal Investigator — Antalya Training and Research Hospital
Locations (1):
- Antalya Training and Research Hospital, Antalya, Muratpaşa, Turkey (Türkiye)